CLINICAL TRIAL: NCT00120393
Title: A Phase IIIB, Open-label, Randomized, Multi-center Study Evaluating the Effect on Serum Lipids Following a Switch to ATV/r in HIV-1 Infected Subjects Who Have Achieved Virologic Suppression on a LPV/r Based Regimen.
Brief Title: Study of HIV Patients With Undetectable Viral Load and Abnormal Lipids Switching to Atazanavir/Ritonavir
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AI424-100
Record Dates: First submitted 2005-07-12; First posted 2005-07-18 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2009-07

CONDITIONS: HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate

ARMS (2):
- G1 (Active Comparator)
  Interventions: Drug: atazanavir/ritonavir +2 NRTIs (immediate Switch Group)
- G2 (Active Comparator)
  Interventions: Drug: LPV/r +2 NRTIs (Delayed/optional Switch Group)

INTERVENTIONS:
Drug: atazanavir/ritonavir +2 NRTIs (immediate Switch Group) — Capsules, Oral, ATV 300mg/RTV 100mg + 2 NRTIs, QD, 48 weeks.
  Other Names: Reyataz
  Arms: G1
Drug: LPV/r +2 NRTIs (Delayed/optional Switch Group) — Capsules, Oral, LPV 400mg/RTV 100mg +2 NRTIs, BID, 24 weeks then option to switch to ATV arm or stay until 48 weeks.
  Arms: G2

SUMMARY:
Patients with HIV who are virologically suppressed on a lopinavir/ritonavir combination highly active antiretroviral therapy (HAART) regimen but with elevated non-HDL cholesterol are randomized to remain on lopinavir/ritonavir or change to atazanavir/ritonavir in combination with current nucleoside reverse transcriptase inhibitors (NRTIs).

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* LPV/RTV-based HAART for at least 6 months
* HIV-1 RNA less than 50c/mL (confirmed)
* Non-HDL higher than 160 mg/dL
* CD4 of at least 50 cells/mL

Exclusion Criteria:

* Use of lipid-lowering agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2004-01; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
To compare the Week 12 percent change from baseline in fasting non-HDL cholesterol between subjects who are switched to an ATV/RTV-containing regimen and those who continue on a LPV/RTV based regimen.

SECONDARY OUTCOMES:
Mean percent change in fasting non-HDL cholesterol at Weeks 24 and 48.
Mean change in cholesterol measures at Weeks 12, 24 and 48.
Mean percent changes from baseline in fasting glucose and insulin at Weeks 12, 24 and 48.
The proportion of subjects receiving lipid lowering therapy at Weeks 24 and 48.
The proportion of subjects with LDL cholesterol less than 130mg/dL at Weeks 12, 24 and 48.
The proportion of subjects with non-HDL cholesterol less than 160mg/dL at Weeks 12, 24 and 48.
The frequency and severity of all clinical and laboratory AEs and discontinue for AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (14):
- United States (12):
  - Local Institution, Phoenix, Arizona
  - Local Institution, Bakersfield, California
  - Local Institution, Los Angeles, California
  - Local Institution, San Francisco, California
  - Local Institution, Miami, Florida
  - Local Institution, Boston, Massachusetts
  - Local Institution, New York, New York
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Portland, Oregon
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Columbia, South Carolina
  - Local Institution, Dallas, Texas
- Canada (2):
  - Local Institution, Hamilton, Ontario
  - Local Institution, Montreal, Quebec